CLINICAL TRIAL: NCT02688790
Title: Pharmacokinetics of a Single-Dose of Dalbavancin in Preterm Neonates to Infants Ages 3 Months With Suspected or Confirmed Bacterial Infection
Brief Title: Study Evaluate the PK Profile of Dalbavancin in Infants and Neonates Patients With Known or Suspected Bacterial Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DAL-PK-02; NCT03617042 (obsolete NCT alias)
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Bacterial Infections
Keywords: Dalbavancin; DALVANCE®; Suspected or Confirmed Bacterial Infection
MeSH Terms: conditions — Bacterial Infections | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): One dose of intravenous dalbavancin infusion 22.5 mg/kg in young infants aged greater than 28 days to 3 months
  Interventions: Drug: Dalbavancin
- Cohort 2 (Experimental): One dose of intravenous dalbavancin infusion 22.5 mg/kg in term neonates (defined as gestational age at or greater than 37 weeks) aged up to 28 days
  Interventions: Drug: Dalbavancin
- Cohort 3 (Experimental): One dose of intravenous dalbavancin infusion 22.5 mg/kg in preterm neonates (defined as gestational age of 32 weeks, up to 37 weeks) aged no more than 28 days
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin
  Other Names: Dalvance®

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetic (PK) profile of a single intravenous (IV) infusion dose of dalbavancin, and to evaluate the safety and tolerability of a single dalbavancin IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female patients who are preterm neonates (gestational age

  ≥32 to <37 weeks, aged ≤28 days), term neonates (gestational age ≥37 weeks, aged ≤28 days) or young infants (aged 28 days to 3 months inclusive) who will be receiving at least 24 hours of appropriate non-investigational intravenous antiinfective treatment other than glycopeptide antibiotics for known or suspected bacterial infections. Patients with urinary tract infections due to Gram-positive organisms may be enrolled
* Each patient's parent(s)/legal guardian(s) must be willing and able to provide a signed and dated written informed consent document indicating that they have been informed of all pertinent aspects of the trial
* Each patient's parent(s)/legal guardian(s) must be willing and able, if patient is discharged from the hospital, to return the patient to the hospital or a designated clinic for scheduled visits, or allow a nurse to come to the patient's home for laboratory tests, PK and other out-patient procedures as required by the protocol
* Patients must be expected to survive with appropriate antibiotic therapy and appropriate supportive care throughout the study
* Sufficient intravenous access (peripheral or central) to receive Investigational Product (IP)
* Patients must have an audiologic assessment within 7 days prior to the investigational product infusion consisting of ear specific hearing testing utilizing distortion product evoked otoacoustic emissions,

Exclusion Criteria:

* 1. Treatment with an investigational drug within 30 days preceding the dose of IP
* Patients who are currently receiving intravenous vancomycin or other glycopeptide antibiotics. Dalbavancin may be administered 8 hours after the last dose of vancomycin. Vancomycin or other glycopeptide antibiotics should not be given during the 7 day period following administration of dalbavancin. If intravenous vancomycin or other glycopeptide use is unavoidable during the 7 day period following administration of dalbavancin, this should be documented as a concomitant medication
* Have aspartate aminotransferase (AST), alanine transaminase (ALT) or total bilirubin level > 3 times upper limit of normal (neonates with elevated total bilirubin could participate if conjugated bilirubin was normal)
* Albumin < half lower limit of normal
* Have received a blood or blood component (eg, red blood cells, fresh frozen plasma, platelets) transfusion during the 24-hour period before dosing
* Have any condition (eg. Septic shock, burns, cystic fibrosis, acute hemodynamic instability including those conditions requiring pressor support) that would make the patient, in the opinion of the Investigator, unsuitable for the study (eg, would place the patient at risk, compromise the quality of the data; or interfere with the absorption, distribution, metabolism or excretion of dalbavancin)
* Patients known to have hypersensitivity to glycopeptides
* Moderate or severe renal impairment defined as serum creatinine ≥2 times the upper limit of normal (× ULN) for age OR urine output <0.5 mL/kg/h (measured over at least 8 hours) OR requirement for dialysis)
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of dalbavancin | Day 1, Day 2, Day 5-9 and Day 24-32
Number of patients experiencing a treatment emergent adverse event | Baseline (Day 1) up to Day 35

SECONDARY OUTCOMES:
Maximum plasma drug concentration (Cmax) | Day 1, Day 2, Day 5-9 and Day 24-32
Area under the plasma concentration versus time curve (AUC) | Day 1, Day 2, Day 5-9 and Day 24-32
Apparent total body clearance (CL) of drug from plasma | Day 1, Day 2, Day 5-9 and Day 24-32
Apparent volume of distribution volume of distribution (V) | Day 1, Day 2, Day 5-9 and Day 24-32
Terminal elimination half-life (T1/2). | Day 1, Day 2, Day 5-9 and Day 24-32

CONTACTS AND LOCATIONS:
Overall Officials: Todd Riccobene, Study Director — Allergan, plc
Locations (5):
- United States (5):
  - Mary Birch Hospital for Women and Newborns, San Diego, California
  - University of California, San Diego, San Diego, California
  - University of Louisville, Louisville, Kentucky
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Duke Medical Center, Durham, North Carolina